CLINICAL TRIAL: NCT06438744
Title: The Role of Thread Embedding Acupuncture for Pain and Quality of Life in Endometriosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Marshellia Setiawan, Medical Doctor, Indonesia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-10-1610
Record Dates: First submitted 2024-05-27; First posted 2024-06-03 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2024-05

CONDITIONS: Endometriosis-related Pain
Keywords: endometriosis; pain; ehp30; acupuncture; thread embedding acupuncture
MeSH Terms: conditions — Endometriosis; Pain | interventions — Tea; Standard of Care

STUDY DESIGN:
Intervention Model Description: One-group pretest-posttest clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): TEA combined with standard therapy
  Interventions: Procedure: Thread embedding acupuncture (TEA) + standard therapy

INTERVENTIONS:
Procedure: Thread embedding acupuncture (TEA) + standard therapy — * TEA : one-time TEA using 30 gauge TEA needle with 30 mm polydioxanone thread at CV3 through CV4, SP6 and ST36 bilaterally
  * Standard therapy : 2 mg dienogest daily for 8 weeks after TEA

SUMMARY:
Endometriosis is a common gynecological problem, with pain as the main problem. Pain can be felt for years, in high intensity, continuous, unpredictable, and disrupts the patient's daily life, thereby reducing the quality of life. Dienogest is a progestin-derived drug, the first line therapy for endometriosis pain. Other therapy options include hormonal, non-hormonal therapy, and surgery, but they have a high risk of side effects and recurrence.

In cases of endometriosis, acupuncture has an analgesic effect, modulates hormones and neurotransmitters, strengthens immune cells, and reduces inflammation, therefore improves quality of life. However, the effectiveness of thread embedding acupuncture for endometriosis pain is still rarely published. This research was conducted to determine the effectiveness of thread embedding acupuncture for pain and quality of life in endometriosis patients.

DETAILED DESCRIPTION:
This study is a one-group pretest-posttest clinical trial. Research subjects will receive a one-time thread embedding acupuncture (TEA) combined with dienogest as standard therapy for 8 weeks. The outcomes assessed will be pain intensity (NRS score) and quality of life score (Endometriosis Health Profile-30 core score) 4 and 8 weeks after receiving TEA combined with standard therapy (posttest), compared with standard therapy alone (pretest).

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-45 years.
2. Subjects diagnosed with endometriosis from laparoscopy, ultrasound, or histopathology.
3. Subjects experience at least one type of pain including pelvic pain, dysmenorrhoea, dyspareunia, dyschezia, or dysuria with a minimum NRS score of 4.
4. The subject has undergone endometriosis therapy with dienogest for at least 1 month but the NRS score is still ≥4.
5. Subjects are willing to follow research procedures and sign the informed consent form.

Exclusion Criteria:

1. Subjects who have wounds, inflammation, infection, lumps, or eczema at the puncture site.
2. Pregnant or breastfeeding women.
3. Subjects with blood clotting disorders or who are taking blood thinning medication.
4. Have a history of diabetes mellitus, malignancy, psychiatric disorders, keloids, allergies to stainless steel or PDO threads.
5. Subjects who received surgical therapy in the last 3 months.
6. Subjects who have been undergoing acupuncture therapy in the last 2 weeks or TEA in the last 6 months.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) score | Before treatment, week 4, week 8
  Pain intensity measurement scale consists of 11 points (0-10). The higher the score, the more severe the pain intensity.
  A score of 0 means there is no pain at all, while a score of 10 means the pain is unbearable.

SECONDARY OUTCOMES:
Endometriosis Health Profile-30 (EHP-30) score | Before treatment, week 4, week 8
  Questionnaire measuring quality of life related to health status, specific for patients with endometriosis. The larger the number, the worse the health status.

CONTACTS AND LOCATIONS:
Overall Officials: Marshellia Setiawan, MD, Study Director — Indonesia University
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No